CLINICAL TRIAL: NCT03881644
Title: Investigation of PACAP38 Induced Headache, Migraine and Flushing in Patients With Migraine
Brief Title: PACAP38 Induced Headache, Migraine and Flushing in Patients With Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Nita Katarina Frifelt Wienholtz, Principal Investigator, Medical Doctor, PhD Student, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MigRosExperiment
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Migraine Without Aura
MeSH Terms: conditions — Migraine without Aura | interventions — Sumatriptan; Sodium Chloride; Pituitary Adenylate Cyclase-Activating Polypeptide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACAP38 + Imigran (Active Comparator): Pituitary adenylate cyclase-activating peptide-38 infusion (10 picomol/kg/min) for 20 mins
  AND
  Imigran infusion (0.4 mg/min) for 10 mins
  Interventions: Drug: Imigran; Other: Pituitary adenylate cyclase-activating peptide-38
- PACAP38 + Isotonic Saline (Placebo Comparator): Pituitary adenylate cyclase-activating peptide-38 infusion (10 picomol/kg/min) for 20 mins
  AND
  Isotonic saline for 10 mins (placebo)
  Interventions: Other: Isotonic Saline; Other: Pituitary adenylate cyclase-activating peptide-38

INTERVENTIONS:
Drug: Imigran — All patients will undergo this intervention on one of two study days
  Other Names: Sumatriptan
  Arms: PACAP38 + Imigran
Other: Isotonic Saline — All patients will undergo this intervention on one of two study days
  Arms: PACAP38 + Isotonic Saline
Other: Pituitary adenylate cyclase-activating peptide-38 — All patients will undergo this intervention on both study days
  Other Names: PACAP38

SUMMARY:
The aim is to investigate the incidence of headache, migraine attacks and flushing after pituitary adenylate cyclase-activating peptide-38 (PACAP38) with and without treatment with sumatriptan in patients with migraine

DETAILED DESCRIPTION:
Pituitary adenylate cyclase-activating peptide-38 (PACAP38) plays a role in migraine pathophysiology. Infusions of PACAP38 can trigger migraine-like attacks in some migraine patients and will induce flushing in all patients. We are investigating whether treatment with sumatriptan has an effect on the PACAP38-induced flushing and on whether headache and migraine is induced.

The purpose of this study is to investigate PACAP38-induced headache and migraine in patients with migraine who have been treated with either sumatriptan or placebo using purpose-developed standardized interview. The study will be conducted with a double-blind, placebo-controlled crossover study design.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of migraine, according to IHS criteria
* weight between 50 - 100 kilograms
* women in fertile age must not be pregnant and must use adequate contraception

Exclusion Criteria:

* migraine more than 5 days per month in average over the past year
* any primary headache other than migraine, apart from tension-type headache which must be less than 5 days per month
* headache < 48 hours before experimental day
* migraine < 72 hours before each experimental day
* daily / frequent use of any medication apart from contraceptive medication
* use of any drug less than 5 times the half-life of the drug at the time of the experiment
* women who are pregnant or breast-feeding at the time of the experiment
* anamnestic or clinical signs of hypertension (systolic blood pressure > 150 mmHg and/or
* diastolic blood pressure > 100 mmHg) or hypotension (systolic blood pressure < 90 mmHg and/or diastolic blood pressure < 50 mmHg)
* anamnestic or clinical signs of mental illness, or abuse of alcohol / drugs
* patients with glaucoma or prostate hyperplasia
* anamnestic or clinical symptoms of any sort that the investigating doctor deemed unfit for participating in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-12-07 (Actual); Study Completion 2019-12-07 (Actual)

PRIMARY OUTCOMES:
Incidence of migraine | From 0 to 12 hours after infusion
  Incidence of migraine after PACAP38-infusion will be estimated through a standardized interview based on the international headache classification for migraine
Effect of Sumatriptan | From 0 to 12 hours after infusion
  Severity of PACAP38-induced headache and migraine after pretreatment with sumatriptan in migraine patients measured by numerical rating scale for pain from 0 ("no pain") to 10 ("worst pain imaginable")

SECONDARY OUTCOMES:
Severity of flushing | From 0 to 4 hours after infusion
  Facial skin blood flow (flushing) will be measured by laser doppler flowmetry to evaluate the severity of PACAP38-induced flushing with and without sumatriptan-treatment
Facial temperature | From 0 to 4 hours after infusion
  PACAP38-induced temperature changes with and without sumatriptan-treatment measured by infrared thermography
Superficial temporal artery diameter | From 0 to 4 hours after infusion
  Superficial temporal artery diameter after PACAP38 with and without sumatriptan-treatment measured by ultrasound
Severity of headache | From 0 to 12 hours after infusion
  Severity of PACAP38-induced headache will be rated on a numerical rating scale for pain from 0 ("no pain") to 10 ("worst pain imaginable")

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, MD,PhD,DMSc, Study Director — Danish Headache Center
Locations (1):
- DanishHC, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wienholtz NKF, Christensen CE, Zhang DG, Coskun H, Ghanizada H, Al-Karagholi MA, Hannibal J, Egeberg A, Thyssen JP, Ashina M. Early treatment with sumatriptan prevents PACAP38-induced migraine: A randomised clinical trial. Cephalalgia. 2021 May;41(6):731-748. doi: 10.1177/0333102420975395. Epub 2021 Feb 10. PMID 33567890